CLINICAL TRIAL: NCT06494683
Title: Efficacy and Safety of Pueraria Lobata Radix As an Adjuvant Treatment for Type 2 Diabetes Mellitus: a Multicenter, Randomized, Double-blinded, Placebo-controlled Trial
Brief Title: Efficacy and Safety of Pueraria Lobata Radix As an Adjuvant Treatment for Type 2 Diabetes Mellitus
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jiangxi University of Traditional Chinese Medicine (Other)
Collaborators: The Affiliated Hospital of Jiangxi University of Traditional Chinese Medicine (Other); The First Affiliated Hospital of Nanchang University (Other)
Responsible Party: Principal Investigator, Xu Zhou, Professor, Jiangxi University of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JCUCM-DIET-01
Record Dates: First submitted 2024-07-02; First posted 2024-07-10 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2024-07

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Pueraria lobata radix; Ge Gen; Type 2 diabetes mellitus; Randomized controlled trial
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — plant extract, Puerariae Radix

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pueraria lobata radix group (Experimental): Pueraria lobata radix will be made into granules.
  Interventions: Drug: Pueraria lobata radix
- Placebo group (Placebo Comparator): The dosage form, specifications and packaging of the placebo will be no different from those of Pueraria lobata radix granules, and the smell and taste will be basically the same.
  Interventions: Drug: Pueraria lobata radix

INTERVENTIONS:
Drug: Pueraria lobata radix — The dose of Pueraria lobata radix granules is one sachet per day, 1.5g per sachet, which equivalent to 15 g of the original herb.
  Other Names: Ge Gen

SUMMARY:
As a dietary herb, pueraria lobata radix (PLR) has been showed to have hypoglycemic effects in animal experiments. However, there is currently a lack of evidence from randomized controlled trials. Therefore, this randomized, double-blind, placebo-controlled trial aims to assess the efficacy and safety of PLR as an adjunctive treatment for type 2 diabetes mellitus (T2DM).

DETAILED DESCRIPTION:
As a dietary herb, pueraria lobata radix (PLR) has been showed to have hypoglycemic effects in animal experiments. However, there is currently a lack of evidence from randomized controlled trials. Therefore, this randomized, double-blind, placebo-controlled trial aims to assess the efficacy and safety of PLR as an adjunctive treatment for type 2 diabetes mellitus (T2DM).

T2DM is the most prevalent chronic metabolic disease. It has been noted in clinical practice that the limitations of conventional treatment methods, such as secondary failure and adverse reactions, continue to pose challenges for patients in managing their blood glucose levels, preventing them from achieving optimal glycemic control goals. Therefore, it is essential to search for more effective and safe complementary medications.

PLR (Chinese name: Ge Gen) is the dried root of the leguminous plant kudzu (Pueraria lobata (Willd.) Ohwi). In China and other East Asian countries, PLR has been widely used to treat metabolic diseases, including T2DM. The chemical components of PLR include isoflavones, triterpenes, saponins, polysaccharides, coumarin compounds, and alkaloids, with isoflavones being the primary active ingredients of PLR. Multiple animal studies have shown that the main active components in isoflavones, such as puerarin, daidzein, and genistein, effectively increase serum insulin concentrations, lower blood glucose levels, and improve insulin resistance in diabetic mice. Puerarin injection has been widely used in China for the treatment of diabetes and its complications.

PLR is classified as a medicinal and edible herb according to Chinese regulations, demonstrating good safety, with no reports of adverse reactions from long-term consumption in practice. However, there is currently a lack of randomized controlled trial evidence on the use of PLR for assisting in glycemic management. Therefore, this study aims to conduct a randomized controlled trial to evaluate the efficacy and safety of daily PLR treatment for adjunctive management of T2DM.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of type 2 diabetes mellitus according to the International Diabetes Guidelines: fasting blood glucose (FBG) ≥ 126 mg/dl (7.0 mmol/l) or 2-hour postprandial blood glucose ≥ 200 mg/dL (11.1 mmol/l), or HbA1c ≥ 6.5% (48 mmol/mol).
2. Age between 18 and 80 years old.
3. Untreated patients or those currently receiving regular anti-diabetic medication therapy, including oral hypoglycemic drugs and insulin, with no restrictions on types or doses.
4. Blood glucose levels not effectively controlled in the three months prior to baseline screening: HbA1c between 6.5% and 10.5%.
5. Willingness to comply with dietary control requirements during the study.
6. Voluntary participation and signing of informed consent form.

Exclusion Criteria:

1. Type 1 diabetes, gestational diabetes, and special types of diabetes.
2. History of diabetic acute complications, including ketoacidosis, hyperosmolar coma, and lactic acidosis.
3. Pregnant or lactating women, or women planning pregnancy.
4. Allergy history to Pueraria lobata radix.
5. Severe dysfunction of vital organs such as heart, liver, and kidney, malignant tumors, or severe mental disorders.
6. Anticipated poor compliance or language communication impairments.
7. Currently participating in other clinical trials.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-07-25 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
HbA1c | Baseline and Week 12
  Changes from baseline in HbA1c levels

SECONDARY OUTCOMES:
HbA1c | Baseline, Week 4 and Week 8
  Changes from baseline in HbA1c levels
HbA1c response rate | Baseline, Week 4, Week 8 and Week 12
  Proportion of patients with HbA1c < 7.0%
Fasting blood glucose | Baseline, Week 4, Week 8 and Week 12
  Changes from baseline in fasting blood glucose levels
Two-hour postprandial glucose | Baseline, Week 4, Week 8 and Week 12
  Changes from baseline in two-hour postprandial glucose levels
Fasting C-peptide | Baseline, Week 4, Week 8 and Week 12
  Changes from baseline in fasting C-peptide levels
Body mass index | Baseline, Week 4, Week 8 and Week 12
  Changes from baseline in body mass index
Total cholesterol | Baseline and Week 12
  Changes from baseline in total cholesterol levels
Triglycerides | Baseline and Week 12
  Changes from baseline in triglycerides levels
High-density lipoprotein cholesterol | Baseline and Week 12
  Changes from baseline in high-density lipoprotein cholesterol levels
Low-density lipoprotein cholesterol | Baseline and Week 12
  Changes from baseline in low-density lipoprotein cholesterol levels
Non-high-density lipoprotein cholesterol | Baseline and Week 12
  Changes from baseline in non-high-density lipoprotein cholesterol levels
Systolic blood pressure | Baseline, Week 4, Week 8 and Week 12
  Changes from baseline in systolic blood pressure
Diastolic blood pressure | Baseline, Week 4, Week 8 and Week 12
  Changes from baseline in diastolic blood pressure
Severity of diabetes symptoms | Baseline, Week 4, Week 8 and Week 12
  Severity of diabetes symptoms will be scored using the Diabetes Symptom Grading Scale in the "Guiding Principles of Clinical Research on New Drugs of Traditional Chinese Medicines".
Diabetes Specific Quality of Life questionnaire scores | Baseline, Week 4, Week 8 and Week 12
  Quality of life will be measured using the Diabetes Specific Quality of Life questionnaire (DSQL).
Hypoglycemic drug dose | Baseline, Week 4, Week 8 and Week 12
  Changes from baseline in hypoglycemic drug dose
Incidence of any adverse events | Baseline, Week 4, Week 8 and Week 12
  An adverse event is defined as any medically induced harm, excluding those due to nature progression of diabetes mellitus.
Incidence of severe adverse events | Baseline, Week 4, Week 8 and Week 12
  Severe adverse events include adverse events that require hospitalization, induce prolonged hospitalization, disability, or impacts on work capacity, are life-threatening, or cause death.
Incidence of treatment-related adverse events | Baseline, Week 4, Week 8 and Week 12
  The causality of treatment and adverse events will be assessed by the Clinical Event Committee.
Incidence of individual adverse events | Baseline, Week 4, Week 8 and Week 12
  The main concern is hypoglycemia and gastrointestinal reactions.

CONTACTS AND LOCATIONS:
Overall Officials: Xu Zhou, M.D, Principal Investigator — Jiangxi University of Traditional Chinese Medicine
Locations (2):
- China (2):
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The Affiliated Hospital of Jiangxi University of Traditional Chinese Medicine, Nanchang, Jiangxi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen J, Wang J, Yuan L, Xue Q, Zhou J, Ye X, Fan Q, Feng R, Li C, Zhang Y, Zhu W, Li Z, Zhou X. Efficacy and safety of Pueraria lobata radix as an adjuvant therapy for type 2 diabetes mellitus: rationale, design and protocol for a randomised controlled trial. BMJ Open. 2025 May 24;15(5):e092050. doi: 10.1136/bmjopen-2024-092050. PMID 40413050